CLINICAL TRIAL: NCT02732470
Title: Effect of Qi Gong Training on Quality of Life in Patients With Systemic Lupus Erythematous (LuQi)
Acronym: LuQi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I15023
Record Dates: First submitted 2016-03-29; First posted 2016-04-08 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematous; Qi Gong; Quality of life
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Qi Gong (Experimental): The effect of Qi Gong training on quality of life in patients with systemic lupus erythematosus
  Interventions: Other: Qi Gong

INTERVENTIONS:
Other: Qi Gong — The aim of this study is to evaluate the effects of Qi Gong on quality if life in patients with Systemic Lupus Erythematosus

SUMMARY:
Systemic Lupus Erythematosus (SLE) is chronic and systemic autoimmune disease that mainly affecting women and leading to organ damages especially skin, joints, kidneys, central nervous system and heart. In SLE, immune system dysfunction leads to autoantibodies, autoreactive T cells and pro-inflammatory cytokines production. These elements will initiate and maintain organ damages. Patients with SLE have disease flares followed by period of remission. Flares can occur because of stress, infections, surgery, pregnancy or ultraviolet exposition. Furthermore the chronic nature of SLE is an important factor of depression in these patients.

Qi Gong is an ancient Chinese practice based on relaxation movements, posture and breathing in order to harmonize the body and mind. This practice improves the general state by reducing fatigue and improving sleep. The beneficial effect of Qi Gong in medicine has been studied in several diseases including cancer, diabetes, arterial hypertension and fibromyalgia. Qi Gong seems interesting in depressed patients but also to reduce stress in healthy subjects.

The aim of this study is to evaluate the effects of Qi Gong on quality if life in patients with SLE. Patients will have two lessons of 60 minutes per week for three months and a collective lesson of 90 minutes per week for three months. The teacher of Qi-Gong will evaluate adherence to the practice of Qi Gong every week. Clinical and biological data will be collected at baseline and at 2th, 4th, 6th, 9th and 12th month. Different evaluation scores and neurotrophin levels will be collected at baseline and at 6th month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Lupus Erythematosus (SLE) according the American Rheumatology Association (ARA) and/or Systemic Lupus International Collaborating Clinics (SLICC) Criteria
* Free and Clarified Consent Term signature.

Exclusion Criteria:

* Patients who have other rheumatologic diseases (rheumatoid arthritis, sjogren syndrome, fibromyalgia, ankylosis spondylitis);
* Systemic Lupus Erythematosus Disease Assessment Index (SLEDAI) > 5;
* Patients with malignancy;
* Patients who do not accept the study rules as time and/or follow-up exercise program time proposed;
* Suspected or pregnancy confirmation;
* Patients with Inability or unwillingness to understand and/or sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Differences in quality of life with the SF-36 Physical Function Domain in patients with SLE at baseline and after a six month practice of Qi-Gong | month 0 - month 6

SECONDARY OUTCOMES:
Quality of life (SF-36), quality of life in patients with SLE | months 0, months 2, months 4, months 9 and months 12